CLINICAL TRIAL: NCT00952146
Title: Transgastric Diagnostic Peritoneoscopy (Laparoscopy) and Appendectomy - A Pilot Study
Brief Title: Transgastric Peritoneoscopy and Appendectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sodra Alvsborgs Hospital (Other)
Collaborators: Borås Lasarett (Other)
Responsible Party: Per-Ola Park, Department of Surgery, South Alvsborg Hospital, Boras, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: South Alvsborg Hospital
Record Dates: First submitted 2009-06-15; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Abdominal Pain
Keywords: NOTES; Transgastric; Appendectomy; Safety; Feasibility
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transgastric peritoneoscopy (Experimental): Only one arm, feasibility study
  Interventions: Procedure: Transgastric peritoneoscopy (NOTES)

INTERVENTIONS:
Procedure: Transgastric peritoneoscopy (NOTES) — Under general anesthesia an endoscope will be passed through the gastric wall into the peritoneal cavity to examine the peritoneal cavity. At the withdrawal of the endoscope, the gastric access in the stomach wall will be closed with T-tags.
  Other Names: No more interventions

SUMMARY:
This study is a feasibility study. Patients with acute abdominal pain who are planning to undergo a diagnostic laparoscopy are asked to participate in the study. The aim of the study is to evaluate if transgastric peritoneoscopy is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute abdominal pain

Exclusion Criteria:

* Patient under 18
* Patient who cannot understand information in Swedish
* Patients previously operated in upper part of the abdomen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To test the feasibility of transgastric peritoneoscopy | When discharged from hospital, 1 month post-op and one year

CONTACTS AND LOCATIONS:
Overall Officials: Per-Ola Park, MD&PhD, Principal Investigator — South Alvsborg Hospital, Boras, Sweden
Locations (1):
- Department of Surgery, South Alvsborg Hospital, Borås, Sweden